CLINICAL TRIAL: NCT07019675
Title: A Phase II, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of SKB518 in Patients With Lung Cancer
Brief Title: A Study of SKB518 in Patients With Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB518-II-02
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — tislelizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2L+ SCLC or non-Squamous NSCLC (Experimental): SKB518 monotherapy
  Interventions: Drug: SKB518
- 2L SCLC (Experimental): SKB518+Tislelizumab or Tislelizumab monotherapy
  Interventions: Drug: SKB518; Drug: Tislelizumab
- 1L ES-SCLC (Experimental): SKB518+Tislelizumab+Carboplatin
  Interventions: Drug: SKB518; Drug: Tislelizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: SKB518 — SKB518 is administered every 3 weeks(Q3W) until radiographic disease progression, intolerable toxicity, or other protocol-specified treatment discontinuation criteria, whichever occurs first.
Drug: Tislelizumab — Tislelizumab is administered every 3 weeks(200 mg, Q3W) until radiographic disease progression, intolerable toxicity, or other protocol-specified treatment discontinuation criteria, whichever occurs first.
  Other Names: Tevimbra
  Arms: 1L ES-SCLC; 2L SCLC
Drug: Carboplatin — Carboplatin is administered at every 3 weeks(AUC 5 mg/mL/min, Q3W) for 4 cycles
  Arms: 1L ES-SCLC

SUMMARY:
This is an open-label, multicenter, phase II study. The purpose of this study is to evaluate the safety, tolerability and preliminary anti-tumor activity of SKB518 in patients with lung cancer. Eligible subjects will receive SKB518 monotherapy, until radiographic disease progression, intolerable toxicity, discontinuation of study treatment required by the subject, or other protocol-specified treatment discontinuation criteria, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old at the time of signing the informed consent form, applicable to both males and females.
2. Non-small cell lung cancer (NSCLC) or small cell lung cancer(SCLC) confirmed by histology or cytology.
3. At least one measurable tumor lesion per RECIST v1.1.
4. Performance status score of 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
5. Expected survival period ≥ 12 weeks.
6. The function of important organs meets the requirements of the protocol.

Exclusion Criteria:

1. Symptomatic or uncontrolled cardiovascular disease
2. History of noninfectious pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD;
3. Subjects with the disease that requires systemic corticosteroid therapy (prednisolone or equivalent dose of similar drugs at a dose of >10 mg/d) or other immunosuppressive therapy within 14 days before the first dose.
4. Human immunodeficiency virus (HIV) positive or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
5. The Investigator considers other situations that will interfere with the evaluation of the study intervention or the safety of the subjects or the interpretation of the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
AE | Up to 24 months
  Incidence and severity of Adverse Events (AEs)
ORR in specific arms | Up to 24 months
  Objective Response Rate (ORR) assessed by the investigators per RECIST v1.1
PFS in specific arm | Up to 24 months
  Progression-Free Survival (PFS) assessed by the investigators per RECIST v1.1

SECONDARY OUTCOMES:
PFS in specific arms | Up to 24 months
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
DOR in specific arms | Up to 24 months
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
OS | Up to 24 months
  Time from start of treatment to death due to any reason.
Pharmacokinetics | Up to 24 months
  Maximum and minimum drug concentrations (Cmax and Cmin) of SKB518-ADC and SKB518-TAb (antibody-drug conjugate and total antibody forms of SKB518) in Serum; Cmax and Cmin of SKB518-Free Payload in Plasma
Immunogenicity | Up to 24 months
  Anti-Drug Antibody(ADA) Titre of SKB518

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Shanghai Pulmonary Hospital (Affiliated to Tongji University), Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin